CLINICAL TRIAL: NCT01989195
Title: Efficacy of EVP 1001-1 (SeeMore) in the Assessment of Myocardial Viability in Patients With Cardiovascular Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Phillip C. Yang, MD, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24224
Record Dates: First submitted 2013-11-12; First posted 2013-11-20 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: ISCHEMIC CARDIOMYOPATHY
Keywords: ISCHEMIC OR CORONARY HEART DISEASE; MYOCARDIAL INFARCTION; MAGNETIC RESONANCE IMAGING; DELAYED GADOLINIUM ENHANCEMENT MRI; MANGANESE-ENHANCED MRI; INFARCT VOLUME/SIZE; ALL CAUSE MORTALITY; VENTRICULAR ARRHYTHMIAS
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CORONARY DISEASE SUBJECT (Experimental): ALL SUBJECTS IN THIS STUDY HAVE PREVIOUSLY DOCUMENTED CORONARY ARTERY DISEASE BY ANGIOGRAPHY
  Interventions: Drug: 'SEEMORE' - MANGANESE-ENHANCED MRI CONTRAST REAGENT

INTERVENTIONS:
Drug: 'SEEMORE' - MANGANESE-ENHANCED MRI CONTRAST REAGENT — EACH SUBJECT UNDERWENT 2 CARDIAC MRI PROCEDURES: ONE WITH MAGNEVIST (GADOLINIUM), ONE WITH SEEMORE (MANGANESE) REAGENT
  * CARDIAC MRI USING STANDARD DOSE OF 0.2mMOL/KG MAGNEVIST IV (IN THE VEIN)
  * CARDIAC MRI USING SEEMORE REAGENT, DOSE: 0.35CC/KG IV (IN THE VEIN) 1 WEEK AFTER GADOLINIUM MRI

SUMMARY:
The investigator hopes to introduce a novel MRI contrast agent with SeeMore ™ that directly defines viable myocardium. Identifying viable myocardium non-invasively using cardiac MRI is still a moving target and a question we plan to answer more definitively with the SeeMore ™ contrast. Though well tested in small and large animals and Phase I & II clinical trials, the investigators would like to determine the efficacy of the SeeMore contrast further in a clinical setting.

SeeMore is a new manganese (Mn)-based intravenous imaging agent being developed to enhance magnetic resonance imaging (MRI). While Mn has long been known to have desirable magnetic and kinetic properties for MRI, use in humans was not initially possible due to cardiovascular depression and electrocardiogram (ECG) changes, including prolongation of PR and QTc intervals, associated with intravenous administration [1-5]. SeeMore provides Mn in a form that maintains the desired magnetic and kinetic properties while overcoming the cardiovascular toxicity of Mn. SeeMore is taken up into heart cells (primarily via addition of calcium to avoid cardiotoxic effects; please refer to US patent #5,980,863). The potential to distinguish healthy heart tissue from unhealthy heart tissue based on a specific sustained pattern of enhancement provides a basis for evaluating the performance of SeeMore in heart patients. It may be possible to enhance the utility of MRI for heart disease through the use of an imaging agent that is specifically taken up into heart cells. SeeMore is the only cardiac-specific agent being developed for this purpose. Unlike nuclear perfusion agents, SeeMore is not radioactive and does not require special handling, shielding, transport or storage. In addition, the specific pattern of enhancement achieved in the heart muscle persists over time, offering potential benefits over the nonspecific extracellular agents currently available for MRI or X-ray/CT procedures. This feature allows full use of the high resolution of MRI, since there is not a trade-off of high spatial resolution for temporal (first-pass) resolution. It is anticipated the features offered by SeeMore along with the high resolution, three dimensional attributes of MRI will result in higher accuracy than is available with other current modalities in practice, including stress echocardiograms, cardiac MRI using gadolinium contrast and nuclear studies such as SPECT and PET. This will be evaluated in this study and serve as the basis for pivotal registration studies.

All components of SeeMore™ are USP and are approved for use as drugs in man, orally and/or intravenously.

DETAILED DESCRIPTION:
This is an open-label, baseline-controlled study. An initial cohort study of patients to conduct safety evaluation will be conducted before proceeding with the additional patients. In this initial cohort, a patient will be dosed based on the Phase 1 and 2 clinical trial data evaluation completed by Eagle Vision Pharmaceutical, Inc.

Starting 30 minutes before the cardiac MRI scan (CMR), the subjects will take a 4 mg tablet of ondansetron by mouth. CMR will subsequently take place and SeeMore™ will then be administered approximately 15 minutes into the scan for contrast enhanced images. SeeMore™ will be administered intravenously over approximately one minute. The subjects will each receive 0.28 mL/kg of SeeMore™. All subjects will be monitored closely from before ondansetron administration until their discharge from the imaging center. If positive delayed-enhanced MRI is detected, the subject will undergo MEMRI within 1 week. The investigators plan to perform imaging with CMR and SeeMore™ within a week after standard gadolinium-based delayed enhanced imaging by CMR (performed as clinically indicated within Stanford Hospital by the patient's physician) to directly compare the two different contrast enhanced images (SeeMore vs Gadolinium in determining viable myocardium).

Parameters to be Measured:

A standard physical examination will be performed within 24 hours prior to dosing and at the end of experimental MEMRI imaging (approximately 1 hour post dosing). A standard 12-lead EKG will be performed both before the experimental MR study and after the experimental MR study to assure no significant EKG changes have occurred. HR will be measured before and after the study. After the study, the patient will have another standard 12-lead EKG performed to compare with the pre-MRI 12-lead EKG. The patient's symptoms will be reassessed 1 hour and 1 year after infusion of the SeeMore contrast. Adverse events (AEs) and discomforts will be recorded until discharge from the imaging center. Any clinically relevant changes from baseline in vital signs, ECG rhythm, clinical chemistries or physical condition and all AEs will be followed until resolution or until the outcome is known. Primary efficacy will be based on determining whether the heart is normal or abnormal and if abnormal whether there is an infarction, ischemia or both. This provides the basis for calculating sensitivity, specificity, accuracy and predictive values. In addition, the location, size, conspicuity and associated confidence for any disease will be recorded.

The study will be stopped for any significant adverse cardiovascular event including cardiovascular death, myocardial infarction, ventricular arrhythmia, ICD firing, congestive heart failure, hospitalization, or syncope.

ELIGIBILITY:
Inclusion Criteria:

-

All subjects to be entered must:

* be at least 18 years of age.
* if female, be nonpregnant as evidenced by a serum pregnancy test and using a medically-approved method of birth control, or post-menopausal or surgically sterile
* provide written informed consent after having received oral and written information about the study
* be in stable health based on medical history, examination and tests

Exclusion Criteria:

- have a positive pregnancy test (females)

* received an investigational drug or device within 30 days prior to administration of SeeMore?
* have known hypersensitivity to ondansetron or other selective serotonin 5HT3 receptor blockers
* have a history of drug abuse or alcoholism
* are taking a digitalis preparation or calcium channel blocker
* have a history of torsades or prolonged QT/QTc interval
* have NYHA Grade IV heart failure
* have abnormal liver function tests or a history of liver disease
* have uncontrolled hypertension (Systolic Blood Pressure > 140 or Diastolic BP > 90 consistently at baseline)
* have abnormal baseline potassium or calcium values or hemoglobin less than 10 g/dl
* are noncompliant or otherwise unlikely to perform as required by the protocol
* have pretest likelihood of CAD for which the requisite number of subjects have been entered
* develop an arrhythmia prior to or during either of the exercise tests; SeeMore? should not be administered.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip C. Yang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CORONARY DISEASE SUBJECT: ALL SUBJECTS IN THIS STUDY HAVE PREVIOUSLY DOCUMENTED CORONARY ARTERY DISEASE BY ANGIOGRAPHY
  'SEEMORE' - MANGANESE-ENHANCED MRI CONTRAST REAGENT: EACH SUBJECT UNDERWENT 2 CARDIAC MRI PROCEDURES: ONE WITH MAGNEVIST (GADOLINIUM), ONE WITH SEEMORE (MANGANESE) REAGENT
  * CARDIAC MRI USING STANDARD DOSE OF 0.2mMOL/KG MAGNEVIST IV (IN THE VEIN)
  * CARDIAC MRI USING SEEMORE REAGENT, DOSE: 0.35CC/KG IV (IN THE VEIN) 1 WEEK AFTER GADOLINIUM MRI
Period: Overall Study
Arm/Group | CORONARY DISEASE SUBJECT
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CORONARY DISEASE SUBJECT
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: COMPARISON OF MYOCARDIAL INFARCTION SIZE MEASUREMENTS USING INVESTIGATIONAL MANGANESE-ENHANCED MRI (MEMRI) OR DELAYED GADOLINIUM ENHANCED MRI (DEMRI)
Description: Measured as percentage of myocardial injury volume to the total left ventricular myocardial volume
Time Frame: Day 1 (1 MRI)
Measure: Mean (Standard Deviation); unit: percentage of infarct to Left Ventricle
Groups:
- DEMRI CORONARY DISEASE SUBJECT: ALL SUBJECTS IN THIS STUDY HAVE PREVIOUSLY DOCUMENTED CORONARY ARTERY DISEASE BY ANGIOGRAPHY
  DEMRI - MAGNEVIST (GADOLINIUM)
  * CARDIAC MRI USING STANDARD DOSE OF 0.2mMOL/KG MAGNEVIST IV (IN THE VEIN)
  * CARDIAC MRI USING SEEMORE REAGENT, DOSE: 0.35CC/KG IV (IN THE VEIN) 1 WEEK AFTER GADOLINIUM MRI
- INVESTIGATIONAL MANGANESE-ENHANCED MRI (MEMRI): ALL SUBJECTS IN THIS STUDY HAVE PREVIOUSLY DOCUMENTED CORONARY ARTERY DISEASE BY ANGIOGRAPHY
  MEMRI- SeeMore
  * CARDIAC MRI USING STANDARD DOSE OF 0.2mMOL/KG MAGNEVIST IV (IN THE VEIN)
  * CARDIAC MRI USING SEEMORE REAGENT, DOSE: 0.35CC/KG IV (IN THE VEIN) 1 WEEK AFTER GADOLINIUM MR
Arm/Group | DEMRI CORONARY DISEASE SUBJECT | INVESTIGATIONAL MANGANESE-ENHANCED MRI (MEMRI)
Number analyzed (Participants) | 6 | 6
percentage of infarct to Left Ventricle | 41 (11.4) | 18.25 (1.7)
Statistical Analysis 1: Comparison: DEMRI CORONARY DISEASE SUBJECT vs INVESTIGATIONAL MANGANESE-ENHANCED MRI (MEMRI); Test type: Superiority or Other; p < .05, t-test, 2 sided

2. Secondary Outcome: SAFETY AND TOLERABILITY OF MANGANESE CONTRAST REAGENT
Description: QRS Duration: SUBJECTS UNDERWENT PRE- AND POST-MRI EKG TESTING TO ASSESS ANY ADVERSE SYMPTOMS OR SIGNS. THE POST EKG WAS PERFORMED AFTER MEMRI SCAN WERE COMPLETE. EKG WAS NOT OBTAINED BEFORE AND AFTER DEMRI.
  Measured the difference in heart rate per EKG before and after MEMRI study.
Time Frame: Pre MRI and Post MRI on same day (Day 1)
Measure: Mean (Standard Deviation); unit: Change in QRS Duration in milliseconds
Arm/Group | CORONARY DISEASE SUBJECT
Number analyzed (Participants) | 6
Change in QRS Duration in milliseconds | 10 (8.12)

3. Secondary Outcome: Significant Cardiovascular Event
Description: Hospitalization and procedures for chest pain, arrhythmias, and all-cause mortality
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- CORONARY DISEASE SUBJECT: ALL SUBJECTS IN THIS STUDY HAVE PREVIOUSLY DOCUMENTED CORONARY ARTERY DISEASE BY ANGIOGRAPHY
  'SEEMORE' - MANGANESE-ENHANCED MRI CONTRAST REAGENT: EACH SUBJECT UNDERWENT 2 CARDIAC MRI PROCEDURES: ONE WITH MAGNEVIST (GADOLINIUM), ONE WITH SEEMORE (MANGANESE) REAGENT
  * CARDIAC MRI USING STANDARD DOSE OF 0.2mMOL/KG MAGNEVIST IV (IN THE VEIN)
  * CARDIAC MRI USING SEEMORE REAGENT, DOSE: 0.35CC/KG IV (IN THE VEIN) 1 WEEK AFTER GADOLINIUM MRI
  Outcome measurement followed for both as all subjects received both MEMRI and DEMRI.
Arm/Group | CORONARY DISEASE SUBJECT
Number analyzed (Participants) | 6
participants | 0

4. Secondary Outcome: Heart Rate: SAFETY AND TOLERABILITY OF MANGANESE CONTRAST REAGENT
Description: SUBJECTS UNDERWENT PRE- AND POST-MRI EKG TESTING TO ASSESS ANY ADVERSE SYMPTOMS OR SIGNS. THE POST EKG WAS PERFORMED AFTER MEMRI SCAN WERE COMPLETE. EKG WAS NOT OBTAINED BEFORE AND AFTER DEMRI.
  Measured the difference in heart rate per EKG before and after MEMRI study.
Time Frame: Pre MRI and Post MRI on same day (Day 1)
Measure: Mean (Standard Deviation); unit: Heart Rate change in beats per minute
Arm/Group | CORONARY DISEASE SUBJECT
Number analyzed (Participants) | 6
Heart Rate change in beats per minute | 7.83 (3.54)

ADVERSE EVENTS:
Groups:
- CORONARY DISEASE SUBJECT: ALL SUBJECTS IN THIS STUDY HAVE PREVIOUSLY DOCUMENTED CORONARY ARTERY DISEASE BY ANGIOGRAPHY
  'SEEMORE' - MANGANESE-ENHANCED MRI CONTRAST REAGENT: EACH SUBJECT UNDERWENT 2 CARDIAC MRI PROCEDURES: ONE WITH CLINICAL MAGNEVIST (GADOLINIUM), ONE WITH EXPERIMENTAL SEEMORE (MANGANESE) REAGENT. ADVERSE EVENTS TRACKED FOR SEEMORE MRI.
  - CARDIAC MRI USING SEEMORE REAGENT, DOSE: 0.35CC/KG IV (IN THE VEIN) 1 WEEK AFTER GADOLINIUM MRI
Arm/Group | CORONARY DISEASE SUBJECT
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CORONARY DISEASE SUBJECT (N=6)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No